CLINICAL TRIAL: NCT07191847
Title: CaraClear, Studying Lens Peptides and Extra Ocular Tissue Managed by ACE Pico Protocol in Tear Film Stability, Tear Volume, and Dry Eye Symptoms Using Stem Cells Fortified Eye Drops
Brief Title: Assessment of CataClear, Tear Film Stability, Tear Volume, and Dry Eye Symptoms Using Stem Cells Fortified Eye Drops
Acronym: CataClear
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ace Cells Lab Limited (Industry)
Collaborators: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCRMED-Cat-002
Record Dates: First submitted 2025-04-21; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Dry Eye; Cataract
Keywords: dryeye; catclear
MeSH Terms: conditions — Dry Eye Syndromes; Cataract | interventions — Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: 2 drops in each eye 3 times daily
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- corneal opacity clearing (Other): selecting the cases of corneal opacity and treat with 2 drops 3 times daily for 12 weeks
  Interventions: Biological: eye drops

INTERVENTIONS:
Biological: eye drops — apply 2 drops 3 times daily for 12 weeks

SUMMARY:
Dry Eye Disease (DED) is a multifactorial condition that affects the ocular surface, leading to discomfort, tear film instability, and potential visual disturbances. Its global prevalence ranges between 5% and 50%, making it a significant cause of reduced quality of life and a growing burden on healthcare systems. Cataract, defined as a progressive opacification of the lens, remains the leading cause of preventable blindness worldwide, responsible for about 33% of all cases, affecting an estimated 94 million people. Its incidence increases with age and is influenced by factors such as ultraviolet exposure, diabetes, smoking, and genetic predisposition. Low- and middle-income countries (LMICs) face a disproportionately high burden due to limited access to surgical care. The economic impact of cataract is profound, including both direct costs (surgery, post-op care) and indirect costs (lost productivity, caregiver dependency), with global productivity losses estimated at $53 billion annually. Beyond economics, cataract significantly impairs quality of life, contributing to psychological distress, depression, loss of independence, and increased risk of cognitive decline. Addressing this burden requires integrated strategies that ensure equitable access to treatment, reduce financial barriers, and include psychosocial support. In parallel, emerging regenerative therapies such as stem cell-fortified eye drops offer new hope. These treatments, utilizing mesenchymal stem cells (MSCs), aim to restore ocular surface health in conditions like DED by reducing inflammation and enhancing tissue repair. The current study evaluates the efficacy of such drops in improving tear film stability, tear volume, and overall clinical symptoms using advanced diagnostic tools.

DETAILED DESCRIPTION:
Dry eye disease (DED) is a multifactorial condition affecting the ocular surface, characterized by symptoms of discomfort, visual disturbances, tear film instability, and potential damage to the ocular surface. DED impacts patients' quality of life and poses a significant healthcare burden, with an estimated global prevalence ranging from 5% to 50%.

Cataract, a progressive opacification of the ocular lens leading to visual impairment, remains the foremost cause of preventable blindness globally, constituting a significant public health burden. According to the World Health Organization (WHO), an estimated 94 million individuals worldwide are affected by cataract-related visual disability, with the condition accounting for approximately 33% of all cases of blindness. The prevalence of cataract exhibits marked demographic and geographic heterogeneity, correlating strongly with advancing age, ultraviolet radiation exposure, metabolic disorders (e.g., diabetes mellitus), tobacco use, and genetic predisposition. While age-related cataracts dominate in populations over 50 years, congenital and traumatic forms contribute to morbidity across all age cohorts. Low- and middle-income countries (LMICs) bear a disproportionate burden, with cataract blindness rates up to threefold higher than in high-income regions due to limited access to surgical interventions and preventive care.

The socioeconomic ramifications of cataract-induced visual impairment are profound. Direct costs, including surgical expenses, postoperative care, and corrective devices, impose substantial financial strain on healthcare systems and households, particularly in resource-limited settings. Indirect costs, such as lost labor productivity, caregiver dependency, and reduced educational attainment, further exacerbate economic disparities. In LMICs, where out-of-pocket expenditures dominate healthcare financing, cost-related barriers delay surgical treatment, perpetuating cycles of disability and poverty. A meta-analysis estimated annual global productivity losses attributable to cataract at $53 billion, underscoring its macroeconomic impact.

Concurrently, cataract-associated visual decline engenders significant psychological morbidity. Patients frequently report diminished quality of life (QoL), characterized by heightened anxiety, depression, and social isolation due to functional limitations in daily activities (e.g., mobility, self-care). The loss of independence, particularly among elderly populations, exacerbates feelings of helplessness and stigmatization. Furthermore, delayed intervention correlates with irreversible neuroadaptive changes in the visual cortex, compounding psychological distress. Emerging evidence also highlights the bidirectional relationship between cataract-related disability and mental health disorders, with untreated visual impairment increasing susceptibility to cognitive decline and dementia.

Addressing the global cataract burden necessitates integrated strategies that combine equitable access to surgical care, cost-reduction initiatives, and psychosocial support systems. Understanding the interplay of epidemiological, economic, and mental health dimensions is critical to mitigating its multisectoral impact on human health and societal well-being.

Emerging therapies, including regenerative approaches like stem cell-fortified eye drops, show promise in addressing underlying pathophysiological mechanisms. These therapies leverage mesenchymal stem cells (MSCs) to promote ocular surface regeneration and repair by modulating inflammation and enhancing tissue healing.

This study aims to evaluate the efficacy of stem cell-fortified eye drops in improving tear film stability, tear volume, and clinical symptoms of DED, utilizing advanced diagnostic technologies for comprehensive assessments.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-80 years.
* Diagnosed with dry eye disease (based on clinical criteria such as OSDI scores and Schirmer test results).

Exclusion Criteria:

* Exclusion Criteria:

  * History of ocular surgery or trauma.
  * Other ocular diseases (e.g., glaucoma, keratitis).
  * Systemic conditions that may interfere with study outcomes (e.g., autoimmune diseases).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Slit-lamp grading + AS-OCT (structural clarity) | 12 weeks
  Assess the therapeutic efficacy of stem cell-fortified eye drops in the corneal opacity

SECONDARY OUTCOMES:
BCVA (functional improvement) | 12 weeks
  detect corneal improvement

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Yasser Sayyed Saif, Prof of ophthalmology, Principal Investigator — Beni-Suef University
Locations (1):
- British center for regenerative medicine, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
1. outcome of the application of the drops with 2 weeks evaluation
  2. any adverse effects
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- See also: Related Info — http://www.ace-cells.co.uk